CLINICAL TRIAL: NCT07407751
Title: Disorders of the Lateral Nasal Wall and Nasal Septum in Patients Candidate for Septorhinoplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mahmoud Mohamed, assisstant lecturer of otorhinolaryngology, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-12-6MD
Record Dates: First submitted 2026-01-16; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Septoplasty Surgeries
MeSH Terms: interventions — Rhinoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with lateral nasal wall disorders (Other): patients with latersl nasal wall disorders such as (middle turbinate hypertrophy, inferior turbinate hypertrophy, concha bullosa, nasal valve collapse) in case inferior turbinate hypertrophy we will do turbinoplasty in case middle turbinate hypertrophy and concha bullosa we will do excision of the medial half of the turbinate in case nasal valve collpase we will manage it using spreader and or batten graft
  Interventions: Procedure: rhinoplasty
- patients with nasal septum disorders (Other): patients with nasal septum disoreders such as ( severe deviated septum either C or S shaped, caudal septum dislocation, fracture cartilagenous septum, maxillary crest deviations, spurred vomer) in severe deviated septum we will do submucous resection of the septum in caudal septum dislocation we will refix the septum to the anterior septal angle in fracture cartilagenous septum we will do septoplasty in maxillary crest deviation we will excise it using ostetomies in spurred vomer we will excise it by bone nippler
  Interventions: Procedure: septoplasty

INTERVENTIONS:
Procedure: rhinoplasty — in case inferior turbinate hypertrophy we will do turbinoplasty in case middle turbinate hypertrophy and concha bullosa we will do excision of the medial half of the turbinate in case nasal valve collpase we will manage it using spreader and or batten graft
  Arms: patients with lateral nasal wall disorders
Procedure: septoplasty — in severe deviated septum we will do submucous resection of the septum in caudal septum dislocation we will refix the septum to the anterior septal angle in fracture cartilagenous septum we will do septoplasty in maxillary crest deviation we will excise it using ostetomies in spurred vomer we will excise it by bone nippler
  Arms: patients with nasal septum disorders

SUMMARY:
Our aim of this study is to provide a detailed description of the lateral nasal wall and nasal septum disorders faced by the surgeon in septorhinoplasty operation and evaluation of therapeutic techniques for their management

DETAILED DESCRIPTION:
Septorhinoplasty is among the most frequently performed plastic surgeries and a common surgical procedure in the field of head and neck. A minor modification of 1 mm can significantly affect the surgical result, necessitating an in-depth understanding of nasal anatomy and adjacent structures on the part of the surgery. The surgical goal for these patients is to address both aesthetic and functional issues, ultimately enhancing their quality of life.

Advancements in understanding the anatomy and physiological characteristics of the nose have paralleled the evolution of surgical remedies for obstructive and aesthetic nasal issues.

The nasal septum carries out several functions, such as splitting the nasal passage into two distinct compartments, maintaining the shape of the nasal dorsum, columella, and nasal tip. Disruptions, be it from injury or innate malformations, in the septum can result in substantial nasal obstruction and visible nasal deformities. The architecture of the nasal septum is composed of distinct osseous and cartilaginous elements, which encompass the perpendicular plate of the ethmoid bone, the vomer bone, and the septal cartilage.

A flawless, undeviated septum ensures that incoming air is humidified, warmed, cleansed, and made appropriate for gas exchanges in the lung alveoli. However, a deviated septum can create various degrees of nasal blockage and modifications in nasal respiration. Disruptions in the airflow can result in olfactory impairment, impairment in the purification and humidification of respiratory air, and diminished oxygen intake. Additionally, anatomical aberrations in the septum can cause epistaxis (nosebleeds), chronic sinusitis, and commonly manifest as visible alterations in the nose's exterior appearance. Septum deviation indicates a departure from the midline, whether of the bone or cartilage, or both.

Common deformities associated with the septum include the subluxation of the rectangular cartilage from the maxillary ridge, or its deviations, which block the nasal floor and distort laminar airflow. Also, Deviation of the caudal portion of the nasal septum may result in nasal obstruction, a crooked nose, and columellar irregularities. The correction of a severely deviated caudal septum is one of the most difficult challenges for the otolaryngologist.

One potential cause of treatment failure may be misidentification of other comorbid causes of nasal obstruction, specifically nasal valve collapse (NVC). Nasal valve collapse not only affects function but also shape of the nose, concurrent NVC is often viewed as an important feature to identify prior to a septorhinoplasty to prevent need for revision surgery .

On each lateral wall of the nasal cavity, there are three bony projections known as nasal turbinates. Disorders in the lateral wall can affect the function of the nose. In a condition known as concha bullosa, the turbinate has a double layer of bone instead of a single layer.

ELIGIBILITY:
Inclusion Criteria:

* All sept rhinoplasty patients aged between 16-60 years

Exclusion Criteria:

1. participants who had a history of major craniofacial trauma or surgeries
2. conditions such as acromegaly or gigantism
3. fungal infections in the paranasal sinuses
4. craniofacial malignancies
5. chronic rhinosinusitis
6. congenital anomalies like cleft lip or cleft palate.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
straight nose | 2 months
  A straight good looking external nasal framework with straight dorsal nose without nasal valve collapse Postoperative standardized frontal and lateral 2D photographs will be rated by 2 independent blinded experts Patient satisfaction will be assessed using FACE-Q rhinoplasty module

SECONDARY OUTCOMES:
Nasal Airway Patency | 1 month
  A straight nasal septum without any deviations or deformities and patent nasal airway without turbinate hypertrophy by endoscopic assessment Airway patency will be assessed by NOSE Score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Eugene Tardy M, Regan Thomas J. Cummings Otolaryngology- Head and Neck Surgery, 5th ed. Mosby: 2015.chapter 36; P.544-508. 2. Aziz T, Ansari K, Lagravere MO, Major MP, Flores- Mir C. Effect of non- surgical maxillary expansion on thenasal septum deviation: a systematic review. Prog Orthod. 2015;16:15. [DOI:10.1186/s40510-015-0084-y] [PMID] [PMCID]. 3. Samrid R, Chaisiwamongkol K, Thanaviratananich S, Sukhorum W, Yimdee J, Iamsaard S. The anatomical study of the nasal septum in north- east Thai Cadavers. Srinagarind Med J. 2013;28(4):279-81. 4. Kenyon G. Nasal Anatomy and Analysis. Otolaryngol Clin An Int J. 2013;5(1):34-42. [DOI:10.5005/aijoc-5-1-12] 5. Bailey BJ, Johnson JT, Newlands SD. (editors). Head & neck surgery-otolaryngology, 4th ed. Philadelphia, Lippincott Williams & Wilkins;2006. 6. Brennan HG, Parkes ML. Septal surgery: the high septal transfixion. Int J Surg. 1973;58(10):732. 7. D'Ascanio L, Manzini M. Quick septoplasty: surgical technique and learning curve. Aesthetic Plast Surg. 2009;33(6):814-8. [DOI:10.1007/s00266-009-9388-y] [PMID] 8. Baumann I, Baumann H. A new classification of septal deviations. Rhinology. 2007;45(3):220-3. 9. Byrd HS, Constantian MB, Guyuron B, Pastorek N. Revision rhinoplasty. Aesthet Surg J. 2007.27(2):175-87. [DOI:10.1016/j.asj.2007.02.001] [PMID] 10. Hong SD, Lee NJ, Cho HJ, Jang MS, Jung TY, Kim HY, Chung SK, Dhong HJ. Predictive factors of subjective outcomes after septoplasty with and without turbinoplasty: can individual perceptual differences of the air passage be a main factor? Int Forum Allergy Rhinol. 2015;5(7):616-21. 11. Becker SS, Dobratz EJ, Stowell N, Barker D, Park SS. Revision septoplasty: review of sources of persistent nasal obstruction. Am J Rhinol. 2008;22(4):440-4.